CLINICAL TRIAL: NCT00510601
Title: LDL Apheresis for the Treatment of Congestive Heart Failure
Brief Title: Treating Congestive Heart Failure Using a Device to Remove Cholesterol
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Patrick Moriarty, MD, FACP, FACC (Other)
Collaborators: Kaneka Medical America LLC (Industry)
Responsible Party: Sponsor-Investigator, Patrick Moriarty, MD, FACP, FACC, Director, Clinical Pharmacology, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10282
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Heart Decompensation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: Kaneka Liposorber

INTERVENTIONS:
Device: Kaneka Liposorber — LDL-apheresis on a bi-weekly basis
  Other Names: Liposorber LA-15 System (Kaneka, Osaka, Japan)

SUMMARY:
A pilot study to examine the effects of LDL-Apheresis on patients with Stage III Congestive Heart Failure.

Study hypothesis: Decreased blood viscosity from receiving LDL-apheresis will decrease workload on the heart and improve symptoms associated with the progression of Congestive Heart Failure

DETAILED DESCRIPTION:
Patients who qualify for the study will receive 7 bi-weekly LDL-Apheresis treatments with the Kaneka Liposorber device. Patients will assess their CHF symptoms using the KC Cardiomyopathy questionnaire prior to each treatment. Blood levels of certain indices related to CHF and safety profile labs will be drawn before and after the first and last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, between the age of 18 and 85 years old. If female, must guarantee that pregnancy will not occur for duration of study
* Presence of Left ventricular systolic dysfunction due to ischemic or non-ischemic cardiomyopathy and have symptoms of New York Heart Association Class III chronic Heart failure (CHF)
* Left ventricular ejection fraction (LVEF) ≤ 35% as measured by radionuclide angiography
* Subject must be on optimal conventional heart failure therapy including Beta-blocker in target or maximally tolerated doses for at least 3 months prior to entry into the study, and/or an angiotension receptor blocker (ARB) for at least 30 days prior to study entry. Subjects on ACE inhibitors, with approval of their physician, have been switched to an ARB one week before initiating apheresis
* Other optimal conventional therapy have been taken for at least 30 days prior to initiation of apheresis
* Subject is able to complete the 6-minute walk test and the Kansas City Congestive Heart Failure Quality of Life Questionnaire (KCCQ)
* Not currently in, or planning to participate in other studies

Exclusion Criteria:

* Age <18 years, or >85 years of age
* Poor venous access
* CHF due to, or associated with, uncorrected primary valvular disease, uncorrected thyroid disease, obstructive/hypertrophic cardiomyopathy, pericardial disease, amyloidosis, active myocarditis, malfunctioning artificial heart valve, uncorrected congenital heart disease, or primary pulmonary hypertension
* Subject has undergone a cardiac revascularization, valvular surgery, or bi-ventricular resynchronization procedure within six months prior to initiation of apheresis treatment
* Subject is listed for transplantation and is expected to be transplanted within 6 months of initiation of apheresis treatment
* Subject has had a myocardial infarction within 6 months prior to initiation of apheresis treatment
* Subject with electrocardiogram (ECG) recorded at initial screening showing particular abnormalities
* Subject has sustained VT, unless precipitated by an event such as an acute myocardial infarction, induction by catheter replacement, or by an electrophysiology procedure, or addressed by placement of an automatic implantable cardiac defibrillator (AICD)
* Subject has an AICD that has fired for any ventricular arrhythmia within 90 days of the initial visit
* Subject has unstable angina
* Subject on a mechanical assist device
* Subject has evidence of concomitant disease that may interfere with the natural course of the subjects underlying heart failure for the duration of the study
* Subject has poorly controlled diabetes mellitus
* Subject is currently taking study prohibited medication
* Subject is unable to tolerate Beta blocker therapy or asthma, has a heart rate of <55 bpm, or the presence of second or third degree heart block without an implanted pacemaker, and first-degree heart block with a PR interval > 220 milliseconds
* Subject has active disease, that in the opinion of the Investigator, may adversely affect the safety and efficacy of the treatment or the life span of the patient
* Subject has history of, or is currently abusing alcohol or illicit drugs
* Subject has serum potassium <4.0 mEq/L or >5.5mEq/L at initial visit
* Subject has serum digoxin level of >1.2ng/mL at time of initial visit
* Subject is pregnant or at risk of becoming pregnant during study
* Subject is currently lactating
* Subject has participated in a clinical drug or device trial in the last 90 days
* Subject has demonstrated noncompliance with previous medical regimens
* Subject is currently hospitalized, and is not hemodynamically stable, or has an acute cardiac or non-cardiac illness that requires further hospitalization
* Subject is unable, or unwilling to change from an ACEI to an ARB
* Subject has a known hypersensitivity to heparin or ethylene oxide
* Subject has a known Low-density lipoprotein cholesterol (LDL-C) level of >130mg/dl

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Improved Symptoms score on KCCQ | 3 Months
Improved Ejection Fraction on ECHO | 3 Months
Improved distance during 6-minute walk test | 3 Months

SECONDARY OUTCOMES:
Various lab measurements measured pre and post the 1st and last treatment, including blood viscosity | Approximately 2 hours, 3 months apart

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Moriarty, M.D., Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States